CLINICAL TRIAL: NCT00717821
Title: A Randomised, Controlled, Open-label, French Multicenter Parallel Group Study to Compare the Maintenance of Haemoglobin Level With Once Monthly Administration of C.E.R.A. (Continuous Erythropoietin Receptor Activator) Versus Epoetin Beta or Darbepoetin Alfa in Patients With Chronic Kidney Disease on Haemodialysis
Brief Title: A Study of Once Monthly Intravenous or Subcutaneous Mircera in Participants With Chronic Kidney Disease on Hemodialysis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21145
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator; epoetin beta; Darbepoetin alfa

ARMS (2):
- Methoxy Polyethylene Glycol-epoetin Beta (Experimental): Participants who are receiving SC or IV epoetin beta or darbepoetin alfa will receive monthly injections of methoxy polyethylene glycol-epoetin beta, with the starting dose of 120 or 200 micrograms calculated from the last weekly dose of epoetin beta or darbepoetin alfa previously administered, using the same route of administration (SC or IV). Thereafter, when the hemoglobin concentration will increase or decrease in a clinically significant amount, a dose adjustment will be performed according to specific provided guidance. Total duration of treatment will be up to 48 weeks.
  Interventions: Drug: Methoxy Polyethylene Glycol-epoetin Beta
- Epoetin Beta or Darbepoetin Alfa (Active Comparator): Participants who are receiving SC or IV epoetin beta or darbepoetin alfa will continue to receive the same treatment (epoetin beta or darbepoetin alfa at the same dose, same administration intervals, and the same route of administration). When necessary, dose adjustments will be performed according to Summary of Product Characteristics (SmPC). Total duration of treatment will be up to 48 weeks.
  Interventions: Drug: Epoetin Beta; Drug: Darbepoetin Alfa

INTERVENTIONS:
Drug: Methoxy Polyethylene Glycol-epoetin Beta — Participants who are receiving SC or IV epoetin beta or darbepoetin alfa will receive monthly injections of methoxy polyethylene glycol-epoetin beta, with the starting dose of 120 or 200 micrograms calculated from the last weekly dose of epoetin beta or darbepoetin alfa previously administered, using the same route of administration (SC or IV). Thereafter, when the hemoglobin concentration will increase or decrease in a clinically significant amount, a dose adjustment will be performed according to specific provided guidance. Total duration of treatment will be up to 48 weeks.
  Other Names: Mircera; C.E.R.A
  Arms: Methoxy Polyethylene Glycol-epoetin Beta
Drug: Epoetin Beta — Participants who are receiving SC or IV epoetin beta will continue to receive the treatment at the same dose, same administration intervals, and the same route of administration. When necessary, dose adjustments will be performed according to SmPC. Total duration of treatment will be up to 48 weeks.
  Arms: Epoetin Beta or Darbepoetin Alfa
Drug: Darbepoetin Alfa — Participants who are receiving SC or IV darbepoetin alfa will continue to receive the treatment at the same dose, same administration intervals, and the same route of administration. When necessary, dose adjustments will be performed according to SmPC. Total duration of treatment will be up to 48 weeks.
  Arms: Epoetin Beta or Darbepoetin Alfa

SUMMARY:
This 2 arm study will compare the hemoglobin maintenance with once monthly methoxy polyethylene glycol-epoetin beta (Mircera) administration versus epoetin beta or darbepoetin alfa in participants with chronic kidney disease on hemodialysis. Participants will be randomized to receive either monthly intravenous (IV) or subcutaneous (SC) methoxy polyethylene glycol-epoetin beta (at a starting dose of 120 or 200 micrograms, calculated from the last weekly dose of epoetin beta or darbepoetin alfa previously administered), or standard therapy (IV or SC epoetin beta once, twice or thrice weekly, or IV or SC darbepoetin alfa once a week or twice a week).

ELIGIBILITY:
Inclusion Criteria:

* regular long term hemodialysis with same schedule for greater than or equal to (>=) 12 weeks
* continuous IV or SC maintenance epoetin beta or darbepoetin alfa therapy, with the same dosing interval during the previous month, and no change in total weekly dose

Exclusion Criteria:

* transfusion of red blood cells during previous 2 months
* significant acute or chronic bleeding
* poorly controlled hypertension requiring hospitalization or interruption of epoetin beta/darbepoetin alfa treatment in previous 6 months
* weekly dose of epoetin beta greater than (>) 16000 international units (IU), or weekly dose of darbepoetin alfa >80 micrograms during previous month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2008-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients maintaining average Hb concentration within target range (10-12g/dL) during evaluation period. | Weeks 16-24

SECONDARY OUTCOMES:
Mean change in Hb concentration between reference and evaluation period, and mean time spent in Hb range of 10-12g/dL during evaluation period. | Weeks 16-24
Dose adjustments, RBC transfusions, AEs. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (80):
- France (80):
  - Abbeville
  - Albi
  - Amilly
  - Angers
  - Annonay
  - Antony
  - Aubagne
  - Aulnay-sous-Bois
  - Avignon
  - Bagnols-sur-Cèze
  - Beauvais
  - Besançon
  - Beuvry
  - Béziers
  - Bois-Bernard
  - Bordeaux
  - Brest
  - Cabestany
  - Caen
  - Cannes
  - Carpentras
  - Castelnau-le-Lez
  - Chamalières
  - Charleville-Mézières
  - Clermont-Ferrand
  - Colmar
  - Compiègne
  - Creil
  - Créteil
  - Dijon
  - Draguignan
  - Évry
  - Fleury-Mérogis
  - Hyères
  - La Chaussée-Saint-Victor
  - La Rochelle
  - La Tronche
  - Le Mans
  - Le Petit-Quevilly
  - Le Port-Marly
  - Lille
  - Lliie
  - Lyon
  - Manosque
  - Marseille
  - Meaux
  - Metz
  - Montpellier
  - Mulhouse
  - Muret
  - Nantes
  - Orléans
  - Paris
  - Perpignan
  - Pessac
  - Pierre-Bénite
  - Poissy
  - Poitiers
  - Quincy-sous-Sénart
  - Reims
  - Rouen
  - Rueil-Malmaison
  - Saint-Benoît
  - Saint-Brieuc
  - Saint-Denis
  - Saint-Maurice
  - Saint-Ouen
  - Saint-Pierre-des-Corps
  - Saint-Priest-en-Jarez
  - Saint-Quentin
  - Saintes
  - Strasbourg
  - Tassin-la-Demi-Lune
  - Toulon
  - Toulouse
  - Trappes
  - Vandœuvre-lès-Nancy
  - Vannes
  - Vienne
  - Villeurbanne

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Locatelli F, Choukroun G, Truman M, Wiggenhauser A, Fliser D. Once-Monthly Continuous Erythropoietin Receptor Activator (C.E.R.A.) in Patients with Hemodialysis-Dependent Chronic Kidney Disease: Pooled Data from Phase III Trials. Adv Ther. 2016 Apr;33(4):610-25. doi: 10.1007/s12325-016-0309-6. Epub 2016 Mar 10. PMID 26965694